# **GEM-1202** (**GRAY-B**)

## STATISTICAL PLAN

Statistical Results Report Version 1.8

November 28, 2013

**TITLE:** Single-group, multicenter Phase II Clinical Trial on the combination of Radiotherapy and Ipilimumab for the treatment of patients with melanoma and brain metastases. (GEM STUDY: RADIATION AND YERVOY IN PATIENTS WITH MELANOMA AND BRAIN METASTASES)

| PROMOTER: GEM Study |
|---------------------|
| STUDY COORDINATOR: |

## **INDEX**

Add headings (Format> Paragraph styles) and they will appear in the index.

## **Tables:**

Add headings (Format> Paragraph Styles) and they will appear in the index.

## Figures:

Add headings (Format> Paragraph Styles) and they will appear in the index.

#### 1. RESULTS

#### 1.1. PATIENTS ASSESSED

#### **POPULATIONS** (following definitions in section 9.2 of the protocol)

- included patients and patients (safety population): Of the <u>58 patients</u> included, all patients were considered within the population of <u>patients treated</u> since allthem had received the minus one dose of Ipilimumab. Baseline characteristics, drug exposure analysis, and safety are presented in this population (n = 58).
- **EVALUABLE PATIENTS:** will include all patients who have received at least one dose of ipilimumab and complete treatment with RTCT.

Table 1. Populations

| Table 1. Fopulations | | |
|--------------------------------------|-------|-------|
| | | N (%) |
| Patients included | Yes | |
| ratients included | Total | |
| Patients treated (Safety Population) | Yes | |
| | Total | |
| | Yes | |
| Evaluable patients | No | |
| | Total | |

Table 2. Evaluable patients for the study according to hospital

| | Table 2. Evaluable patients for the study according to hospital | | | |
|---|---|---|---|---|
| | | No | Yes | Total |
| | | N (%) | N (%) | N (%) |
| Hospital | | | | |

#### Table 3. List of NON-evaluable

| patients<br>Patient | Hospital | RDT Total number<br>duration of Ipilimumab<br>cycles | Reason not evaluable / excluded |
|---|---|---|---|

#### 1.2. BASELINE CHARACTERISTICS

The database was closed on XX-XX-XXXX and based on the population of  $\overline{XX}$  patients included / treated in the study, the baseline characteristics are presented:

Table 4. Baseline characteristics (I)

| | N | Mean (SD | Median (Min-Max) |
|-------------------------------------|---|----------|------------------|
| Age (years) | | | |
| Karnofsky functional status (0-100) | | | |
| Barthel index (0-20) | | | |

| Table 5. Baseline characteristics (II) | | |
|----------------------------------------|---------------|--------|
| | | N (%¹) |
| | Male | |
| Sex — | Female | |
| _ | Total | |
| | 70-80 | |
| <u></u> | 90-100 | |
| KPS — | Not specified | |
| _ | Total | |
| | <15 | |
| Barthel Index | 15-20 | |
| _ | Total | |
| | Mutated | |
| Status B-Raf (Current | Native | |
| Melanoma) | Not specified | |
| _ | Total | |
| | 0 | |
| NIO of lines of muscieus two two or | 1 | |
| N° of lines of previous treatment— | >1 | |
| _ | Total | |
| | Mu tado | |
| Status B-Raf (Previous | Native | |
| Melanoma) | Not specified | |
| • | <br>Total | |
| | Multiple | |
| D 144 | Single | |
| Brain M1 — | Not specified | |
| _ | Total | |
| | 1 | |
| _ | 2 | |
| No. of organs with metastatic | 3 | |
| disease | 4 | |
| _ | 5 | |
| _ | Total | |
| No. of organs with metastatic | ≤2 | |
| disease | > 2 | |
| | Total | |
| Dunin materials | Yes | |
| Brain metastases — | Total | |
| | No | |
| Pulmonary metastases | Yes | |
| • | Total | |
| | No | |
| Hepatic metastases | Yes | |
| | Total | |

| | No |
|-------------------------------|-------|
| Metastasis Skin | Yes |
| | Total |
| | No |
| Gastrointestinal metastases | Yes |
| _ | Total |
| Locoregional lymph node | No |
| metastases - | Yes |
| Hietastases | Total |
| | No |
| Distant lymph node metastases | Yes |
| | Total |

<sup>1:%</sup> with respect to *included patients* with available data.

Table 6. Use of previous BRAF inhibitors

| | | · | N (%¹) |
|---|---|---|---|
| Lice of provious | | No | |
| Use of previous - BRAF inhibitors - | | Yes | |
| DIVAL IIIIIDILOIS - | Total | | |
| | | BRAFi | |
| Type of treatment lin | oo DDAE inhibitor | BRAFi + MEKi | |
| Type of treatment lines BRAF inhibitor | Vemurafenib + Pembrolizumab | | |
| | | Total | |

<sup>1:%</sup> with respect to *included patients* with available data.

Table 7. Corticosteroids at baseline and / or cycle 1

| | | <b>,</b> |
|------------------------------------|-------|----------|
| | | N (%¹) |
| Corticosteroids at baseline and /- | No | |
| or C1 | Yes | |
| 01 01 | Total | |

<sup>1:%</sup> with respect to *included patients* with available data.

Table 8. Mean daily dose (dexamethasone reference)

| | N | Mean (SD | Median (Min-Max) |
|---|---|---|---|
| Mean daily dose (Dexamethasone) | | | |
| 1:% with respect to the patients include | <b>d</b> with ava | ailable data (pa | tients who received |
| corticosteroids and for whom the dose) | | | |

Table 9.: Hematology

| | N | Mean (SD | Median (Min-Max) |
|------------------------------------|---|----------|------------------|
| Leukocytes x10 ^ 3 / uL | | | |
| Eosinophils | | | |
| Baseline laboratory testsBasophils | | | |
| Monocytes | | | |
| Neutrophils | | | |
| Lymphocytes | | | |
| Neutrophils Total x10 ^ 3 / uL | | | |
| Eosinophils Total x10 ^ 3 / uL | | | |
| Basophils Total x10 ^ 3 / uL | | | |
| Total Monocytes x10 ^ 3 / uL | | | |
| Total Lymphocytes x10 ^ 3 / uL | | | |
| Hemoglobin g / dl | | | |
| Platelets x10 ^ 3 / uL | | | |
| Neutrophil / Lymphocyte Ratio | | | |

The mean baseline LDH value was 420.3 U / L.Baseline blood tests

Table 10.: Biochemistry

| | N | Mean (SD | Median (Min-Max) |
|----------------------------------|---|----------|------------------|
| Creatinine (mg / dl) | | | |
| Creatinine Clearance (ml / min) | | | |
| SGOT / AST (U / L) | | | |
| SGTP / ALT (U / L) | | | |
| Total Bilirubin (mg / dL) | | | |
| CRP | | | |
| Ureic Nitrogen or Urea (mg / dL) | | | |
| Glucose (mg / dL) | | | |
| Sodium (mmol / L) | | | |
| Chloride (mmol / L) | | | |
| Bicarbonate (mmol / L) | | | |
| Baseline LDH (U / L) | | _ | |

Table 11. LDH categorized

| | · III Gatogonizoa | |
|----------------------|-------------------|--------|
| | | N (%1) |
| | No | |
| Value of LDH> ULN | Yes | |
| | Total | |
| | No | |
| LDH value> 1.5 * ULN | Yes | |
| | Total | |

<sup>1:%</sup> with respect to *included patients* with available data.

Table 12. Baseline analysis: Endocrine

| | N | Mean (SD | Median (Min-Max) |
|---------------------|---|----------|------------------|
| Cortisol (ug / dl) | | | |
| ACTH (pg / mL) | | | |
| T4 (ug / mL) | | | |
| T3 (ug / mL) | | | |
| TSH (uIU / mL) | | | |
| Prolactin (ng / ml) | | | |

#### 1.3. TREATMENT EXPOSURE

Table 13. IPI treatment (I)

| | 1 | N (%) |
|-----------------------------------|-------|-------|
| | 1 | |
| | 2 | |
| Total number of Ipilimumab cycles | 3 | |
| | 4 | |
| | Total | |
| | Total | |
| | 0 | |
| | 1 | _ |
| number of omissions | 2 | |
| number of offissions | 3 | |
| | Total | |
| | Total | |
| | 0 | |
| | 1 | |
| | 2 | |
| number of reductions | 3 | |
| | 4 | |
| | Total | |
| | Total | |
| | 0 | |
| | 1 | |
| number of delays | 2 | |
| | 3 | |
| | Total | |

1:% with respect to *patients included* with available data

Table 14. RDT treatment (I)

| | | N (%) |
|--------------------|-------|-------|
| Premature end of — | No | |
| RDT ——— | Yes | |
| KDI | Total | |
| | | N (%) |
| Reason for | | |
| interruption of | | |
| RDT treatment | | |

1:% with respect to patients included with available data

Table 15. Duration of RDT

| | N | Mean (SD | Median (Min-Max) |
|------------------------|---|----------|------------------|
| <b>Duration of RDT</b> | | | |

Table 16. Patients with no end date of RDT

| | Patient code | Duration RDT | EndRDT | date ofStart date of RDT |
|---|--------------|--------------|--------|--------------------------|
| 1 | | | | |

#### 1.4. Screening of all patients

median follow-up for  $\underline{the\ patient\ population\ treated}$ , n = XX, was XXmonths.

Table 17. Time tracking all patients

| | N | Mean (SD) | median<br>(Me n-Max) |
|---|---|---|---|
| Follow-up time (months from 1st cycle of Ipilimumab) | | | |

#### 1.5. EFFECTIVENESS ANALYSIS

Following the protocol, the population ofwas used for the efficacy analysis evaluable patients: n = XX (see section 1.1)

#### 1.5.1. OVERALL SURVIVAL (Evaluable)

Survival Overall (OS) is presented for evaluable patients (n = XX). The estimated overall survival at one year (calculated using Kaplan-Meier) was X% (with a 95% CI: XX%) with a median OS of X months (95% CI XX months).

Table 18. Overall survival (evaluable)

| Estimated overall survival | N events | N at risk | % of patients without death | 95% CI | % with death |
|---|---|---|---|---|---|
| at 6 months | | | | | |
| to 12 months | | | | | |
| | N (%) | Median | Min-Max | Standard<br>Error | 95% Confidence interval |
| Overall survival Estimated | | | | | |

Table 19. Overall survival: Events and OS at 1 year (Evaluable)

| | and the state of t | <u> </u> |
|---|---|---|
| | | N (%; 95% CI) |
| | Live | |
| Overall survival | Exitus | |
| | Total | |
| | No | |
| OS at 1 year ( <i>crude</i> ) | Yes | |
| OS at 1 year (crude) | No follow-up at 1 year (or death) | |
| | Total | |
| OS at 1 year ( <i>gross</i> ) (excluding | No | |
| patients with follow-up <1 year and | Yes | |
| without previous death) | Total | |

Figure 1. Estimated overall survival (Evaluable)

Table 20. Time to Exitus (only in patients with death)

| | N | Mean (SD) | Median<br>( Min-Max) |
|----------------|---|-----------|----------------------|
| Time to Exitus | | | |

Table 21. Reasons for leaving the study (evaluable)

| | N (%) |
|------------------|-------|
| Reason<br>Exitus | |

#### 1.5.1.1. OS RATE AT 1 YEAR vs BASAL CHARACTERISTICS

A univariate and multivariate analysis of the possible association between baseline characteristics and the rate was presented below. of global survival per year, using logistic regression models taking death per year as an event.

Table 22. Univariate analysis: 1-year OS rate vscharacteristics baseline

| Table 22. Univariate analysis: 1-year OS rate vscharacteristics baseline | | | | | | |
|---|---|---|---|---|---|---|
| | | | 1-yearOS | | Univariate logistic | regression |
| | | No (death)<br>N (%) | Yes (alive)<br>N (%) | Total<br>N (%) | OR (95% CI) | p -value |
| Age categorized _ | <66 years | | | | | |
| according to | ≥66 years | | | | | |
| median (66 years) | Total | | | | | |
| | Female | | | | | |
| Sex | Male | | | | | |
| | Total | | | | | |
| | 90-100 | | | | | |
| KPS | 70-80 | | | | | |
| | Total | | | | | |
| | 15-20 | | | | | |
| Barthel Index | <15 | | | | | |
| | Total | | | | | |
| Status B-Raf _ | Native | | | | | |
| (Current | Mutated | | | | | |
| Melanoma) | Total | | | | | |
| | > 1 | | | | | |
| No. of lines of | 1 | | | | | |
| previous –<br>treatment _ | 0 | | | | | |
| _ | Total | | | | | |
| Status B-Raf | Native | | | | | |
| (previous | Mutated | | | | | |
| Melanoma) | Total | | | | | |
| | brain Single | | | | | |
| Type of locations – M1 Current – | Multiple | | | | | |
| - | Total | | | | | |
| | No | | | | | |
| Location M1 = Current liver = | Yes | | | | | |
| | Total | | | | | |
| Corticosteroids at | No | | | | | |
| baseline and / or | Yes | | | | | |
| C1 - | Total | | | | | |
| | 1 | | | | | |
| No. of organs _ | 2 | | | | | |
| with metastatic | 3 | | | | | |
| disease | 4 | | | | | |

| | Total |
|----------------------------|--------------------------------|
| No. of organs | ≤2 |
| with metastatic | > 2 |
| disease | Total |
| Neutrop<br>Lymphocyte | ohil /Ratio<br>e(quantitative) |
| Neutrophil /ratio | No |
| Lymphocyte> 3 | Yes |
| (high risk) | Total |
| D DDAE | No |
| Previous BRAF<br>Inhibitor | Yes |
| | Total |
| CRP | value |
| Hemogl | obin value |
| LDH | value |
| | No |
| LDH value> ULN | Yes |
| | Total |
| I Dil values 4.5 * | No |
| LDH value> 1.5 * ULN | Yes |
| 52 | Total |

## 1.5.1.2. 1-YEAR OS RATE vs BASAL CHARACTERISTICS. MULTIVARIATE ANALYSISBaseline

Table 23. Multivariate analysis: 1-year OS rate vscharacteristics

| | Table 23. Wulliva | iliale alialysis. 1-yeal Oo | rate vacilaracteriation | ·3 |
|---|---|---|---|---|
| | | | Multivariate logis | stic regression |
| | | $N^1$ | OR (95% CI) | p-value |
| VVVV | No | | | |
| XXXXX | Yes | | | |
| Constant | | | | |

<sup>1:</sup> patients for whom no data were available are excluded from the model data in all variables included in the multivariate model (n = X).

In the table below, the variables that were not significant have been excluded:

Table 24. Multivariate analysis: 1-year OS rate vscharacteristics<sup>2</sup>

| | terrainate amanger | <b>,</b> | | |
|---|---|---|---|---|
| | | | Multivariate logistic | regression |
| | | N¹ | OR (95% CI) | p-value |
| BaselineXXXXXI - | No | | | |
| Daseille AAAAA – | Yes | | | |

<sup>1:</sup> patients for whom data were not available on all variables included in the multivariate model (n = X) are excluded from the model.

Table 25. Multivariate analysis: 1-year OS rate vscharacteristics baseline

| | | | Multivariate logistic | regression |
|----------|-----|----|-----------------------|------------|
| | | N¹ | OR (95% CI) | p-value |
| XXX | No | | | |
| *** | Yes | | | |
| Constant | | | | |

<sup>1:</sup> patients for whom no data was available in all variables included in the multivariate model (n = X).

## 1.5.1.3. 1-YEAR SG RATE vs BASAL CHARACTERISTICS. MULTIVARIATE ANALYSIS. GOODNESS OF FIT

Table 26. Goodness of fit: Hosmer-Lemeshow

| | Chi-square test | Degrees of freedom | p-value |
|--------------------------|-----------------|--------------------|---------|
| Hosmer and Lemeshow Test | | | |

Table 27. Goodness of fit: Classification table

| | | | Predicted | |
|--------------|-------------|------------|--------------|-----------|
| | | | OS at 1 year | |
| Obse | erved | No (death) | Yes (alive ) | % correct |
| | No (death) | | | _ |
| OS at 1 year | Yes (alive) | | | |

<sup>2: &</sup>lt;u>IMPORTANT NOTE</u>: Those variables that were not significant but that were used for the construction of the multivariate model shown in thetable are not shown in the table *previous*.

| | % Total | | |
|-----|----------------|---------------------|----------------|
| | Table 28. Good | ness of fit: Area ເ | under thecurve |
| AUC | Standard error | p-value | 95% CI |

Figure 2. Goodness of fit: ROC curve

#### 1.5.2. PROGRESSION-FREE SURVIVAL (Evaluables)

## Following the protocol, the population ofwas used for the efficacy analysis evaluable patients: n = X (see section 1.1)

According to protocol: PFS is defined in each patient as the time between the date of the first dose of ipilimumab and the date on which progression is determined or death occurs, whichever occurs first. If a patient dies without prior notification of progression, progression will be considered to have occurred on the date of death. For a patient who undergoes tumor resection during the study, the PFS will be censored on the date of the last tumor evaluation prior to resection. In the case of patients who remain alive and do not show progression, the PFS will be censored on the date of the last tumor evaluation. For patients in whom PE has been determined before week 12 and a subsequent evaluation of EE, PR, or CR is obtained, the date of PE after response (if available) will be used in the analysis. of the SLP; otherwise, these patients will be censored on the date of their last tumor evaluation.

Table 29. Progression-free survival (evaluable)

| - Iu | oic zo. i logic | <u> </u> | i vivai (cvaiaabic) | | |
|---|---|---|---|---|---|
| Estimated progression-free survival | N events | N at risk | % of patients without progression | 95% CI | with progression |
| at 6 months | | | | | |
| to 12 months | | | | | |
| | N (%) | Median | Min-Max | Standard<br>Error | Confidence interval 95% |
| Estimated progression-free survival | | | | | |

Table 30. Progression-free survival and PFS at 6 months (Evaluable)

| Table con 1 togicocien necesar | Trai and Tro at o months (E | - varaubioj |
|---|---|---|
| | | N (%; 95% CI) |
| | Alive (without PE) | |
| Progression free curvival | PE | |
| Progression-free survival | Exitus (without prior PE) | |
| | Total | |
| | No | |
| | Yes | |
| PFS at 6 months (crude) | No follow-up at 6 months | |
| | (or PE before 6m) | |
| | Total | · |
| PFS at 6 months (crude) | No | |
| (excluding patients with follow-up <6 months | Yes | |
| and no PE / previous death) | Total | |

Figure 3. Survival free of Estimated progression (Evaluable)

Table 31. Time to PE (only in patients with PE)

| | N | Mean (SD) | Median<br>(Min-Max) |
|---|---|---|---|
| Time to PFS (months from 1st cycle of Ipilimumab) (only patients with PE) | | | |

#### 1.5.2.1. PFS RATE A 6 MONTHS vs BASAL CHARACTERISTICS

Next, a univariate and multivariate analysis was proposed. e the possible association between the baseline characteristics and the 6-month progression-free survival rate, using logistic regression models taking PD or death as an event at 6-month follow-up.

A univariate analysis was carried out in which none of the following variables showed a statistically significant association (p <0.1) with PFS at 6 months of follow-up and therefore multivariate analysis was not carried out.

Table 32. Univariate analysis: PFS rate at 6m vs Baselinecharacteristics

| | Table 32. Univariate analysis: PFS rate at 6m vs Baselinecharacteristics | | | | | |
|---|---|---|---|---|---|---|
| | | | PFSat 6m | | Univariate logistic | regression |
| | | No (without<br>PD or death)<br>N (%) | Yes (living without PD) N (%) | Total<br>N (%) | OR (95% CI) | p-value |
| Age categorized _ | <66 years | | | | | |
| according to | ≥66 years | | | | | |
| median (66 years) | Total | | | | | |
| | Female | | | | | |
| Sex | Male | | | | | |
| | Total | | | | | |
| | 90-100 | | | | | |
| KPS | 70-80 | | | | | |
| | Total | | | | | |
| | 15-20 | | | | | |
| Barthel Index | <15 | | | | | |
| | Total | | | | | |
| Status B-Raf | Native | | | | | |
| (Current | Mutated | | | | | |
| Melanoma) | Total | | | | | |
| | 0 | | | | | |
| No. of lines of previous | 1 | | | | | |
| treatment _ | >1 | | | | | |
| | Total | | | | | |
| Status B-Raf | Native | | | | | |
| (previous | Mutated | | | | | |
| Melanoma) | Total | | | | | |
| | Single | | | | | |
| Type of locations M1 Current Brain | Multiple | | | | | |
| | Total | | | | | |
| | No | | | | | |
| Location M1 Current liver | Yes | | | | | |
| | Total | | | | | |
| Corticosteroids at_ | No | | | | | |
| baseline and / or | Yes | | | | | |
| C1 | Total | | | | | |

| | 4 |
|----------------------------|-----------------------------|
| | 1 |
| No. of organs | 2 |
| with metastatic | 3 |
| disease | 4 |
| | Total |
| No. of organs | ≤2 |
| with metastatic | > 2 |
| disease | Total |
| | rophil /<br>e(quantitative) |
| RatioNeutrophil | No |
| /Ratio<br>Lymphocyte> 3 | Yes |
| (high risk) | Total |
| Dravious DDAF | No |
| Previous BRAF<br>Inhibitor | Yes |
| | Total |
| CRF | Pvalue |
| Hemogl | obinvalue |
| LDH valu | eLDH value |
| | No |
| > ULN | Yes |
| | Total |
| | No |
| LDH value> 1.5 * ULN | Yes |
| ULN | Total |

Table 33 Multivariate analysis: PFS rate at 6m vs Baseline characteristics

| Table 33 Multivariate analysis. 11 3 rate at only vs baseline characteristics | | | | |
|---|---|---|---|---|
| | | | Multivariate logistic regression | |
| | | N <sup>1</sup> | OR (95% CI) | p-value |
| xxxxx | No | | | |
| | Yes | | | |
| XXXXX | No | | | |
| ^^^^ | Yes | | | |
| Constant | | | | |

<sup>1:</sup> patients for whom data were not available in all variables included in the multivariate model (n = X).

#### 1.5.3. BEST RESPONSE (Evaluable)

Following the protocol, for the efficacy analysis the population ofwas used evaluable patients: n = X (see section 1.1)

Table 34. Best response (Evaluable)

| | | N (%; 95% CI) |
|---|---|---|
| | CR | |
| Post reapones (Criteria modified | PR | |
| Best response (Criteria modified from WHO) | EE | |
| IIOIII WHO) | PE | |
| | NE (Not evaluated) | |
| | Total | |
| | RCri | |
| Best response (Response Criteria | RPri | |
| related to immunity. CRri) | EERI | |
| | PEri | |
| | NEri (Not evaluated) | |
| | Total | |

#### According to protocol: Overall best response rate (TMRG)

The MRG is defined by a population subgroup as the total number of patients treated in the subgroup whose MRG is CR or PR, divided by the total number of patients treated in the subgroup.

Table 35. TMRG (Evaluables)

| | | N (%; 95% CI) |
|-------------------------------------|---------------|---------------|
| | No | |
| TMRG: CR or PR (Modified WHO | Yes | |
| Criteria) | Not evaluated | |
| | Total | |
| | No | |
| TMRG: CR or PR (Response | Yes | |
| Criteria related to immunity. CRri) | Not evaluated | |
| | Total | |

#### According to protocol: Disease control rate (TBI)

TBI is defined as the total number of patients treated in each subgroup whose GRM is CR, PR or EE, divided by the total number of patients treated in the subgroup.

Table 36. TBI (Evaluable)

| | Table Co. 1DI (Evaluabl | N (%; 95% CI) |
|------------------------------------|-------------------------|---------------|
| | No | (11), 1111 17 |
| TCE: CR or PR or EE (Modified | Yes | |
| WHO Criteria) | Not evaluated | |
| | Total | |
| | No | |
| TCE: CR or PR or EE (Response | Yes | |
| Criteria related to immunity. CRri | Not evaluated | |
| | Total | |

Table 37. Time to best response (evaluable)

| | N <sup>1</sup> | Mean (SD) | Median<br>(Min-Max) |
|---|---|---|---|
| Time to best WHO response (months from 1st | | | |
| cycle of ipilimumab) | | | |
| Time to best response CRri (months from 1st | | | |
| cycle of ipilimumab) | | | |

<sup>1:</sup> Patients with response recorded in CRDe

Table 38. Time to best response (Evaluable) according to MRG

| Time to | best response | N¹ | Mean (SD) | Median<br>(Min-Max) |
|---|---|---|---|---|
| | CR | | | |
| Best global response (modified | PR | | | |
| WHO criteria ) | EE | | | |
| | PE | | | |
| Time to | best response | N¹ | Mean (SD) | Median<br>(Min-Max) |
| | RCri | | | |
| Best Overall response (Response RPri | | | | |
| zeet e terum respense (reseptine | C 1XI II | | | |
| Criteria related to immunity. CRri | | | | |

<sup>1:</sup> Patients with response recorded in CRDe

#### According to protocol: Duration of response

The duration of a patient's response is defined as the time elapsed between the date on which the measurement criteria for an overall response of PR or CR are first met (whichever response is recorded first, and if confirmed later) and the date of disease progression or death, whichever comes first. For patients undergoing tumor resection during the study, the duration of response will be censored on the date of the last tumor evaluation prior to resection. In the case of patients who remain alive and do not show progression, the duration of the response will be censored on the date of the last tumor evaluation.

Table 39. Duration of response (Evaluable)

| | N¹ | Mean (SD) | Median<br>(Min-Max) |
|---|---|---|---|
| Duration of response (modified WHO criteria), | | | |
| months | | | |
| Duration of response (Response Criteria related to | | | |
| immunity. CRri) , months | | | |

<sup>1:</sup> Patients with response recorded in CRDe

#### According to protocol: Duration of Stable Disease

The duration of stable disease is defined in patients whose MRG is EE as the time that elapses between the moment when the disease was documented for the first time. EE and date of PE or death (whichever occurs first). In the case of a patient who undergoes tumor resection after week 12 but before disease progression occurs, the duration of stable disease will be censored on the date of the last evaluable tumor evaluation prior to resection. In patients with an EE MRG at week 12, the date of PE after this time (if available) will be used in the analysis of the duration of stable disease. In patients with an EE MRG who have not shown subsequent progression and remain alive, the duration of stable disease will be censored on the date of the last evaluable tumor evaluation.

Table 40. Duration of stable disease (Evaluable)

| 4 | () | |
|----------------|------------|----------|
| N <sup>1</sup> | Mean (SD) | Median |
| | Wican (OD) | Miculaii |

| | (Min-Max) |
|------------------------------------------------------------|-----------|
| Duration of stable disease (modified WHO criteria), months | |
| Duration of stable disease (Response Criteria related to | |
| immunity . CRri), months | |

<sup>1:</sup> Patients with response recorded in CRDe

#### 1.5.4. GRAPHIC REPRESENTATIONS RESPONSE (Evaluable)

Following the researcher's instructions, different graphic representations have been elaborated to evaluate the results of the response (WHO).

Figure 4. Spider plot: Absolute change in the measurements of the lesions with respect to baseline

Figure 6. Waterflow plot: Absolute change in the measurements of the lesions with respect to baseline (according to the use of corticosteroids)

Figure 7. Waterflow plot: Absolute change in the measurements of the lesions with respect to baseline (excluding extreme value) (according to the use of corticosteroids)

Figure 8. Waterflow plot:% change in the measurements of the lesions with respect to baseline (according to the use of corticosteroids)

Figure 9. Waterflow plot:% change in the measurements of lesions with respect to baseline (according to use of corticosteroids) cut by 200%

Figure 10. Waterflow plot:% change in the measurements of lesions with respect to baseline (excluding extreme value) (according to use of corticosteroids)

Figure 11. Waterflow plot:% change in lesion measurements with respect to baseline (according to response)

Figure 12. Waterflow plot:% change in lesion measurements with respect to baseline (excluding extreme value) (according to answer)

Figure 13. Swimmerplot: follow-up Entity of each patient with corticosteroids, response and status at the end of follow-up

#### 1.6. TOXICITIES (Treatment-related AEs)

As specified in the protocol for this analysis, was used the population of treated patients, n = XX.

Table 41. Toxicities

| | | N (%1; 95% CI) |
|--------------------------------------------|--------------|----------------|
| Patients with at least one toxicity, any | No | |
| grade | Yes | |
| grade | Total | |
| | No | |
| Patients with at least one gradetoxicity≥3 | Yes | |
| | Total | |
| | No | |
| Patients with grade 3 toxicities | Yes | |
| | Total | |
| | No | |
| Patients with grade toxicities 4 | Yes | |
| | Total | |
| Patients with grade 5 toxicities | No | |
| Fatients with grade 3 toxicities | Total | |
| | None | |
| | 1 toxicity | |
| No. of gradetoxicities≥3per patient¹ | 2 toxicities | |
| | 3 toxicities | |
| | 4 toxicities | |
| | Total | |

<sup>1:</sup> Patients could present more than one toxicity of the same grade

Table 42. Time between initiation of treatment and toxicity (days)

| | Mean (SD) | Median<br>(Min-Max) |
|---|---|---|
| Time between initiation of treatment and toxicity (days) | | |

The frequencies of toxicities with grade ≥3 are shown below.

Table 43. Toxicities with grade ≥3

| Type of Toxicity | Grade 3<br>N (% <sup>1</sup> ) | Grade 4<br>N (%¹) |
|------------------|--------------------------------|-------------------|

<sup>1:%</sup> calculated with respect to the total number of patients evaluable for safety (n = XX)

Below is a list of the toxicities with grade≥3 per patient with their characteristics.

Table 44. List of grade ≥3 toxicities (patients may present more than one toxicity)

| Patient code | Toxicity and Grade | SAE | Relationship<br>with treatment | Start | date AE End<br>date AE |
|---|---|---|---|---|---|

The most frequent toxicities with their degrees and in ANNEX I : LIST OF TOXICITIES A list of all toxicities is presented.

Table 45. Most frequent toxicities (> 10% on = 5) and their grade

| | | -, 3 |
|------|----------|-------|
| | | N (%) |
| XXXX | Absence | |
| **** | Presence | |
| XXXX | Absence | |
| **** | Presence | |

Table 46. Median time between initiation of treatment and toxicity in the most frequent toxicities (days)

| \ <b>j</b> -/ | |
|---|---|
| | Time between initiation of treatment and toxicity |
| Type of toxicity (most frequent) | Median (days) |

Table 47. Median time between the start of treatment and toxicity in the most frequent toxicities (days) as a function of the MRG rate

| | (days) as a re | inction of the mixo rate | |
|---|---|---|---|
| | Type of Toxicity | Rate of best global<br>response TMRG (PR or<br>CR) (modified WHO<br>criteria) | Median (days) |
| | | No | |
| | XXXX | Yes | |
| | | Total | |
| Adverse Event | | No | |
| | xxxx | Yes | |
| | **** | Not evaluated | |
| | | Total | |

## 1.7. AEs As specified in the protocol for this analysis, was used the population of treated patients, n = XX.

Table 48 AFs

| Table 4 | 017(20 | N. (0/10E0/ OD |
|---|---|---|
| | | N (% <sup>1</sup> 95% CI) |
| | No | |
| Patients with at the least one AE, any grad | e Yes | |
| | Total | |
| | No | |
| Patients with at the least one AE grade≥3 | Yes | |
| | Total | |
| | No | |
| Patients with AEs grade 3 | Yes | |
| | Total | |
| | No | |
| Patients with AEs grade 4 | Yes | |
| | Total | |
| Patients with Grade 5 AEs | No | |
| ratients with Grade 3 ALS | Total | |
| | None | |
| | 1 AE | |
| | 2 AEs | |
| No. of GradeAEs≥3per patient¹ | 3 AEs | |
| to. of GradeAES23per patient | 4 AEs | |
| | 5 AEs | |
| | 11 AEs | |
| | Total | |

<sup>1:</sup> Patients could present more than one AE of the same grade

. present the frequencies of AEs with grade ≥3.

Table 49.with grade ≥3

| AEType of AE | Grade 3<br>N (%¹) | Grade 4<br>N (%¹) |
|--------------|-------------------|-------------------|

<sup>1:%</sup> calculated with respect to the total number of patients evaluable for safety (n = XX)

Table 50. Time between start of treatment and AE

| | Mean (SD) | Median<br>(Min-Max) |
|---|---|---|
| Time between initiation of treatment and AE | • | |

Below are the most frequent AEs with their grades and in ANNEX II: LIST OF ALL AEsAEs a list of allis presented.

Table 51. AEs most frequent (> 10% or= 5) and its grade

| | | nN (%) |
|------|----------|------------|
| XXXX | Absence | 49 (84.5%) |
| ^^^ | Presence | 9 (15.5%) |
| XXXX | Absence | 43 (74.1%) |
| ^^^ | Presence | 15 (25.9%) |

#### 1.8. **SAE**

#### ALL / Related

As specified in the protocol, was used for this analysis the treated patient population,  $n = XX_{...}$ 

Table 52, SAEs

| | Table 32. SALS | |
|------------------|----------------|----------------|
| | | N (%¹; 95% CI) |
| | No | |
| At least one SAE | Yes | |
| | Total | |

1:% with respect to *included patients* with available data.

The SAEs with their details are presented below:

Table 53. List of SAEs with details

| | | idalo coi zioi oi oi tali dotalio | | | |
|---|---|---|---|---|---|
| Relationsl<br>ip with AE<br>treatment | E No. Patient | SAE and grade | Specify<br>relationship<br>AE | Start | date AE End<br>date AE |
| No | 1<br>2<br>3 | | | | |
| Yes | 1<br>2<br>3 | | | | |

The following are the frequencies of SAEs not related to grade ≥3.

Table 54. Unrelated SAEs with grade ≥3

| 14010 0 11 0 111 0 1410 4 07 (20 11111 9 1440 20 | | |
|---|---|---|
| Type of unrelated SAE | Grade 3<br>N (%¹) | Grade 4<br>N (%¹) |

<sup>1:%</sup> with respect to *included patients* with available data.

Below are the frequencies of unrelated SAEs of any grade.

Table 55. List of unrelated SAEsunrelated

| Type of SAE | N (%1) |
|-------------|--------|

<sup>1:%</sup> with respect to *included patients* with available data.

#### **1.9. DEATHS**

As specified in the protocol for this analysis, the treated patient population, n = XX, was used. Deaths in the study or within 30 days after the last dose: ALL / drug related

Table 56. Deaths during the study

| Table of Boatile dailing the stady | |
|---|---|
| | N (%¹; 95% CI) |
| Deaths during the study or within 30 days after the last | No (Exitus but considered out of study) |
| | Yes |
| dose | Not applicable (no death) |
| dose | Total |

1:% regarding the *patients included* with available data.

#### Table 57.list

| Tubio of mot | | | | | | | |
|---|---|---|---|---|---|---|---|
| ExitusExitus during the<br>study or in the 30 days<br>after the last dose | No. | Patient code | Exitus reason Exitus | reason other | Date of last<br>Ipilimumab cycle | Date Exitus | OS time (months since 1st ipilimumab cycle) |
| No | 1 | | | | | | |
| (exitus considered out of | 2 | | | | | | |
| study) | 3 | | | | | | |
| | 1 | | | | | | |
| Yes | 2 | | | | | | |
| | 3 | | | | | | |

#### 2. ANNEXES

#### 2.1. ANNEX I: TOXICITY LIST

The frequencies of all the toxicities listed in the DB are detailed below.

#### Table 58. List of all toxicities

| | Toxicities | N (%) |
|-------|------------|-------|
| Total | | |

#### 2.2. ANNEX II: LIST OF ALL AEs

Below frequencies of all AEs collected in the DB are detailed (toxicities included).

#### Table 59. List of all AEs

| | AEs | N (%) |
|-------|-----|-------|
| Total | | |